CLINICAL TRIAL: NCT04008290
Title: The Effect of Liraglutide on MMC Activity, Gastrointestinal Hormones, Hunger Ratings and ad Libitum Food Intake in Healthy Volunteers
Brief Title: The Effect of Liraglutide on the GIT
Acronym: LIRHV
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: S61865
Record Dates: First submitted 2019-06-11; First posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Obesity
Keywords: Liraglutide; MMC; Motilin; Ghrelin; Hunger; glucose; ad libitum food intake
MeSH Terms: conditions — Obesity | interventions — Liraglutide; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0.6 mg Liraglutide (Experimental): For a duration of 5 consecutive days, subjects will receive a subcutaneous injection in the abdomen of 100 µl containing 0.6 mg liraglutide.
  Interventions: Drug: 0.6 mg Liraglutide
- Placebo (Placebo Comparator): For a duration of 5 consecutive days, subjects will receive a subcutaneous injection in the abdomen of 100 µl saline (0.9%) solution.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 0.6 mg Liraglutide — For a duration of 5 consecutive days, subjects will receive a subcutaneous injection in the abdomen of 0.6 mg liraglutide. The injection will be placed by a trained nurse at 8 o'clock every morning. A wash out period of at least one week will be respected between the two treatment weeks.
  Other Names: Victoza
  Arms: 0.6 mg Liraglutide
Drug: Placebo — For a duration of 5 consecutive days, subjects will receive a subcutaneous injection in the abdomen of placebo (0.9% saline solution). The injection will be placed by a trained nurse at 8 o'clock every morning. A wash out period of at least one week will be respected between the two treatment weeks.
  Other Names: saline solution
  Arms: Placebo

SUMMARY:
Liraglutide is a glucose-like peptide 1 agonist, currently used as an effective weight-loss treatment. Its mechanism of action has not yet been elucidated. We want to investigate whether liraglutide affects MMC activity, gastrointestinal hormone release, glucose whole blood levels, hunger ratings and ad libitum food intake in healthy volunteers.

DETAILED DESCRIPTION:
Liraglutide is a glucose-like peptide 1 (GLP-1) agonist, currently used as an effective weight-loss treatment. Its mechanism of action has not yet been elucidated. GLP-1 infusion in humans suppresses hunger-inducing MMC contractility.

Therefore, we will recruit 15 healthy subjects which will participate to this double-blind, placebo-controlled crossover trial. The subjects will receive both treatment arms: 5 consecutive days of placebo injection or 0.6 mg liraglutide injection. On the 4th day, the injection will be combined with a motility study (fasted state), and on the 5th day with an ad libitum buffet.

The primary outcome of this study is to investigate whether liraglutide decreases MMC activity, measured by a solid-state, high-resolution manometry catheter (only on 4th day of the treatment arm). The amount and preference for certain types of food is tested during an ad libitum free choice buffet (only on 5th day of treatment arm). The effect on gastrointestinal hormone release will be measured by taking blood samples at regular time points (both 4th and 5th day of treatment arm). In parallel with the blood sample collection, glucose whole blood levels are measured. Hunger-related sensations are scored on a visual analog scale of 100 mm at regular time points (both 4th and 5th day of treatment arm).

ELIGIBILITY:
Inclusion Criteria:

* Subject is female or male between 18 and 65 years of age.
* Subject has a BMI between 18 and 25 kg/m² and has a stable body weight for at least 3 consecutive months at the start of the study and keeps a stable weight during the study visits.
* Women of child-bearing potential agree to apply during the entire duration of the trial a highly effective method of birth control, which is defined as those which result in a low failure rate (i.e., less than 1% per year) when used constantly and correctly such as implants, injectables, combined oral contraceptive method, or some intrauterine devices (IUDs), sexual abstinence, or vasectomized partner. Women of nonchildbearing potential may be included if surgically sterile (tubal ligation or hysterectomy) or postmenopausal with at least 2 year without spontaneous menses.
* Subject understands the study procedures and agrees to participate in the study by giving written informed consent.

Exclusion Criteria:

* Subject is under age of legal consent, pregnant or breastfeeding.
* Subject with a BMI ≤ 18 kg/m² or BMI ≥ 25 kg/m².
* Subject has current symptoms or a history of gastrointestinal or other significant somatic or psychiatric diseases or drug allergies.
* Subject has diabetes.
* Subject has a significant heart, lung, liver or kidney disease.
* Subject has any history of a neurological disorder.
* Subject has a history of abdominal surgery. Those having undergone a simple appendectomy more than 1 year prior to the screening visit may participate.
* Subject shows abnormal eating behavior or has an eating disorder.
* History or current use of drugs that can affect glycaemia, gastrointestinal function, motility or sensitivity or gastric acidity.
* History or current use of centrally acting medication, including antidepressants, antipsychotics and/or benzodiazepines (in the last year before screening visit).
* Subject consumes excessive amounts of alcohol, defined as >14 units per week for women and >21 units per week for men.
* Subject is currently (defined as within approximately 1 year of the screening visit) a regular or irregular user (including "recreational use") of any illicit drugs (including marijuana) or has a history of drug (including alcohol) abuse. Further, patient is unwilling to refrain from the use of drugs during this study.
* High caffeine intake (> 500 ml coffee daily or equivalent).
* Inability or unwillingness to perform all of the study procedures, or the subject is considered unsuitable in any way by the principal investigator.
* Recent participation (<30 days) or simultaneous participation in another clinical study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
MMC activity compared between placebo and treatment with liraglutide | The catheter will be placed 1 hour before the subcutaneous administration. Antroduodenal contractility will be measured for 5 hours after liraglutide or placebo injection.
  On the 4th day of a treatment arm, the liraglutide or placebo injection is combined with a motility study. A solid-state, high-resolution manometry catheter is placed to measure intragastric pressure (IGP; mmHg). Antroduodenal contractility will be measured during the fasted state.

SECONDARY OUTCOMES:
Gastrointestinal hormone release compared between placebo and treatment with liraglutide | Reference sample is taken at 7:50 in the morning. Other blood samples are taken from every 30 min after the injection (8am). The 4th day, this stops at 13:00 and the 5th day at 15:00. No samples are taken during the buffet at day 5 (13:30 until 14:15).
  On the 4th and 5th day of a treatment arm, blood samples are taken to measure motilin and ghrelin release in the plasma at regular time points.
Hunger sensations compared between placebo and treatment with liraglutide | Hunger is scored every 5 min for 6 hours at day 4 of the treatment, starting at 7:00 and ending at 13:00. At day 5, hunger is scored every 5 min for 7 hours and 20 min starting at 7:40 and ending at 15:00, except during 13:30 and 14:15 (buffet).
  On the 4th and 5th day of a treatment arm, hunger sensations (hunger, prospective hunger and satiety) are scored on a visual analog scale of 100 mm.
Ad libitum food intake compared between placebo and treatment with liraglutide | The buffet will be given 5 hours after the consumption of a standardized breakfast which was given half an hour after the subcutaneous injection. Subjects have 45 min to finish the buffet.
  On the 5th day of a treatment arm, the liraglutide or placebo injection is combined with an ad libitum buffet test. In the morning, the subjects eat a standardized breakfast. Five hours later, the subjects have the opportunity to eat ad libitum from a free choice buffet. All types of food are presented, and all are weighted before and after the experiment to measure the consumed amount of calories.
Glucose whole blood levels compared between placebo and treatment with liraglutide | Reference sample is taken at 7:50 in the morning. Other glucose samples are taken from every 30 min after the injection (8am). The 4th day, this stops at 13:00 and the 5th day at 15:00. No samples are taken during the buffet at day 5 (13:30 until 14:15).
  On the 4th and 5th day of a treatment arm, glucose whole blood levels are measured directly with a glucometer in parallel with the collection of blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, Principal Investigator — UZ Leuven